CLINICAL TRIAL: NCT02776176
Title: A Prospective Multi-center Randomized Controlled Clinical Trials of Enhanced Recovery After Surgery in Hirschsprung Disease.
Brief Title: Enhanced Recovery After Surgery In Hirschsprung Disease
Acronym: ERASIHD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Weibing Tang (Other)
Collaborators: Xuzhou Medical University (Other); Soochow University (Other); Wuxi People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Weibing Tang, Dr. Weibing Tang, Nanjing Children's Hospital
Organization: Nanjing Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WTang
Record Dates: First submitted 2016-05-15; First posted 2016-05-18 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Hirschsprung Disease
Keywords: enhanced recovery after surgery; hirschsprung disease
MeSH Terms: conditions — Hirschsprung Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ERAS group (Experimental): Patients receive the Enhanced Recovery After Surgery program during the peri-operative period.
  Interventions: Procedure: Enhanced Recovery After Surgery Program
- Traditional group (Other): Patients receive the Traditional program during the peri-operative period.
  Interventions: Procedure: Traditional Program

INTERVENTIONS:
Procedure: Enhanced Recovery After Surgery Program — optimized peri-operative protocol
  Other Names: Fast Track Surgery
  Arms: ERAS group
Procedure: Traditional Program — traditional standard protocol
  Arms: Traditional group

SUMMARY:
The study is designed to determine if enhanced recovery after surgery (ERAS) principles could provide benefit for pediatric patients undergoing radical surgery for Hirschsprung's Disease (HD). Half of patients will receive the ERAS program, while the other half will receive the traditional program.

DETAILED DESCRIPTION:
Optimized peri-operative care within an enhanced recovery after surgery (ERAS) protocol is designed to reduce morbidity after surgery, resulting in a shorter hospital stay. The present study evaluated this approach in the context of radical surgery for pediatric patients with Hirschsprung's Disease(HD). Patients undergoing radical surgery for HD will be enrolled in a randomized clinical trial comparing ERAS protocol vs a control group that received standard care. The primary outcome is median length of postoperative hospital stay. The second outcomes include postoperative complications rates，gastrointestinal function recovery time，mean cost per patient，readmission rates within postoperative 30 days，and the levels of stress and inflammation marker.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Hirschsprung Disease

Exclusion Criteria:

* with other disease
* receive emergency surgery
* need to do the ostomy
* full colonic Hirschsprung Disease

Max Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
median length of postoperative hospital day | 30days

SECONDARY OUTCOMES:
postoperative complications rates | within 30 days
gastrointestinal functional recovery time | within 30 days
mean cost per patient | within 30 days
the readmission rates | within 30 days
the level of stress and inflammation marker | within 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Tang, MD&PhD, Study Chair — Nanjing Children's Hospital Affiliated to Nanjing Medical University
Locations (3):
- China (3):
  - The Children's Hospital Of Soochow University, Suzhou, Jiangsu
  - Wuxi Children's Hospital Affiliated to Wuxi People's Hospital Group, Wuxi, Jiangsu
  - Xuzhou CHildren's Hospital Affilated to Xuzhou Medical College, Xuzhou, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kehlet H, Dahl JB. Anaesthesia, surgery, and challenges in postoperative recovery. Lancet. 2003 Dec 6;362(9399):1921-8. doi: 10.1016/S0140-6736(03)14966-5. PMID 14667752
- [Background] Kehlet H. Enhanced Recovery After Surgery (ERAS): good for now, but what about the future? Can J Anaesth. 2015 Feb;62(2):99-104. doi: 10.1007/s12630-014-0261-3. Epub 2014 Nov 13. No abstract available. PMID 25391731
- [Background] Bakker N, Cakir H, Doodeman HJ, Houdijk AP. Eight years of experience with Enhanced Recovery After Surgery in patients with colon cancer: Impact of measures to improve adherence. Surgery. 2015 Jun;157(6):1130-6. doi: 10.1016/j.surg.2015.01.016. Epub 2015 Mar 16. PMID 25791027
- [Background] Nygren J, Hausel J, Kehlet H, Revhaug A, Lassen K, Dejong C, Andersen J, von Meyenfeldt M, Ljungqvist O, Fearon KC. A comparison in five European Centres of case mix, clinical management and outcomes following either conventional or fast-track perioperative care in colorectal surgery. Clin Nutr. 2005 Jun;24(3):455-61. doi: 10.1016/j.clnu.2005.02.003. Epub 2005 Apr 9. PMID 15896433
- [Background] King PM, Blazeby JM, Ewings P, Franks PJ, Longman RJ, Kendrick AH, Kipling RM, Kennedy RH. Randomized clinical trial comparing laparoscopic and open surgery for colorectal cancer within an enhanced recovery programme. Br J Surg. 2006 Mar;93(3):300-8. doi: 10.1002/bjs.5216. PMID 16363014
- [Background] Lassen K, Coolsen MM, Slim K, Carli F, de Aguilar-Nascimento JE, Schafer M, Parks RW, Fearon KC, Lobo DN, Demartines N, Braga M, Ljungqvist O, Dejong CH; ERAS(R) Society; European Society for Clinical Nutrition and Metabolism; International Association for Surgical Metabolism and Nutrition. Guidelines for perioperative care for pancreaticoduodenectomy: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):817-30. doi: 10.1016/j.clnu.2012.08.011. Epub 2012 Sep 26. PMID 23079762
- [Background] Nygren J, Thacker J, Carli F, Fearon KC, Norderval S, Lobo DN, Ljungqvist O, Soop M, Ramirez J; Enhanced Recovery After Surgery Society. Guidelines for perioperative care in elective rectal/pelvic surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):801-16. doi: 10.1016/j.clnu.2012.08.012. Epub 2012 Sep 26. PMID 23062720
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, MacFie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery Society. Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Clin Nutr. 2012 Dec;31(6):783-800. doi: 10.1016/j.clnu.2012.08.013. Epub 2012 Sep 28. PMID 23099039
- [Background] Mortensen K, Nilsson M, Slim K, Schafer M, Mariette C, Braga M, Carli F, Demartines N, Griffin SM, Lassen K; Enhanced Recovery After Surgery (ERAS(R)) Group. Consensus guidelines for enhanced recovery after gastrectomy: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Br J Surg. 2014 Sep;101(10):1209-29. doi: 10.1002/bjs.9582. Epub 2014 Jul 21. PMID 25047143
- [Derived] Tang J, Liu X, Ma T, Lv X, Jiang W, Zhang J, Lu C, Chen H, Li W, Li H, Xie H, Du C, Geng Q, Feng J, Tang W. Application of enhanced recovery after surgery during the perioperative period in infants with Hirschsprung's disease - A multi-center randomized clinical trial. Clin Nutr. 2020 Jul;39(7):2062-2069. doi: 10.1016/j.clnu.2019.10.001. Epub 2019 Oct 16. PMID 31676258
- [Derived] Lu C, Xie H, Li H, Geng Q, Chen H, Mo X, Tang W. Feasibility and efficacy of home rectal irrigation in neonates and early infancy with Hirschsprung disease. Pediatr Surg Int. 2019 Nov;35(11):1245-1253. doi: 10.1007/s00383-019-04552-8. Epub 2019 Sep 18. PMID 31535199